CLINICAL TRIAL: NCT02373709
Title: Sequence Variations of Genes in the Estrogen Pathway and Perinatal Depression
Status: Active, not recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/539/F
Record Dates: First submitted 2015-02-22; First posted 2015-02-27 (Estimated); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Postnatal Depression; Genetic Predisposition
MeSH Terms: conditions — Depression, Postpartum; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva samples for DNA extraction
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: Perinatal depression: Cases will be defined as those with a depressive episode with onset during the antenatal or postnatal period.
- Controls: No perinatal depression: Controls will be defined as those who score < 7 on Edinburgh Postnatal Depression Scale and/or no episode of clinical depression from pregnancy until 6 months postnatal.

SUMMARY:
To elucidate the disease pathway of perinatal depression by identifying genetic variants which could play a role in predisposing to the condition and/or lead to better understanding of the pathogenesis of the condition. This is achieved by investigating for associations between oestrogen receptor genetic variants and perinatal depression.

DETAILED DESCRIPTION:
Perinatal (antenatal and postnatal) depression is a common complication of childbearing, affecting 10 to 20% of mothers. In general, women are exposed to fluctuations in estrogen level during childbearing years, especially during pregnancy and following childbirth. For a subgroup of women with genetic predisposition rendering them more sensitive to such changes, pregnancy or childbirth can act as a trigger for the onset of perinatal depression.

A case control study will be conducted to evaluate the association of variants in estrogen receptor and related genes with the disorder in our population. Women attending antenatal and postnatal clinics will be screened with the Edinburgh Postnatal Depression Scale and cases will be identified. DNA from controls who are well throughout the antenatal and postpartum period and cases meeting DSM IV criteria for depressive disorder will be genotyped for various genetic variants. The distribution of single nucleotide polymorphisms and haplotypes and non-genetic risk factors will be compared between cases and controls and within the case group. The risk factors for postnatal depression in relation to peripartum factors such as demographic, obstetric, anaesthetic and pain outcomes will be investigated.

As perinatal depression is known to contribute to inadequate self-care and poor compliance with prenatal care, early diagnosis and treatment interventions are critical for the health and well-being of both mother and infant. In the short term, identified genetic markers that increase vulnerability to puerperal triggering of depression can be an additional screening tool to identify at-risk expectant mothers for early management during a very critical period for mother, infant, and family. In the long run, it may lead to identification of new pathways or treatment targets for this common but under-studied disorder.

ELIGIBILITY:
Inclusion Criteria:

* Anthropometric profile: age 21-35 years; Chinese race; Chinese ancestry for all 4 grandparents
* Natural conception (not artificially assisted)
* Cases: depressive episode during antenatal period or < 6 months postnatal at time of recruitment; patients with past diagnosis of depression must have been well for 3 months before pregnancy
* Controls: well during antenatal period or > 6 months postnatal at time of recruitment; no family history of depression or affective disorders

Exclusion Criteria:

* Other psychiatric disorders (non-mood disorders) namely schizophrenia and substance dependence
* Previously diagnosed neurological disorders

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Chinese women attending antenatal and postnatal clinics in KK Women's and Children's Hospital and National University Hospital, Singapore.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2010-10; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Perinatal depression | Antenatal and postnatal period
  Defined as meeting Diagnostic and Statistical Manual for Psychiatric Disorders, Fourth Edition (DSM-IV) criteria for major depression through an interview by a clinician using Structured Clinical Interview for Diagnosis (SCID).

CONTACTS AND LOCATIONS:
Overall Officials: Ene Choo Tan, Ph.D., Principal Investigator — KK Research Centre
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore